CLINICAL TRIAL: NCT00790062
Title: Comparison of the Effectiveness of 3 Different Dose Regimens of Oxytocin in Preventing Uterine Atony and Postpartum Hemorrhage During Vaginal Delivery
Brief Title: Oxytocin Regimen to Prevent Atony and Postpartum Hemorrhage During Vaginal Delivery: 3-arm RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alan Tita, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: F070910007; 5K12HD001258-09 (NIH)
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Uterine Atony; Postpartum Hemorrhage
Keywords: Uterine atony; Postpartum hemorrhage; clinical trial; Prophylactic oxytocin
MeSH Terms: conditions — Uterine Inertia; Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxytocin 10 units/500cc (Active Comparator): 1 dose only for prophylaxis given over 1 hour
  Interventions: Drug: Oxytocin
- Oxytocin 40 units/500cc (Experimental): One dose only given over 1 hour. Per DSMB recommendations, this intermediate arm was stopped Jan 2010.
  Interventions: Drug: Oxytocin
- Oxytocin 80U/500cc (Experimental): 1 dose only given over 1 hour
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — See arms
  Other Names: Pitocin

SUMMARY:
This is a double-blind 3-arm randomized clinical trial to determine whether higher dose oxytocin regimens (compared to the standard regimen) reduce the frequency of uterine atony and postpartum hemorrhage after vaginal delivery. Uterine atony is a loss of tone in the uterine musculature which can cause acute postpartum hemorrhage, which is the major cause of maternal mortality worldwide. Oxytocin is routinely administered postpartum in the US and effectively reduces uterine atony. The optimal dose of oxytocin for vaginal delivery is not known.

DETAILED DESCRIPTION:
Same as brief summary. Prospective interim monitoring (stopping) rules will be assessed upon recruitment of 2/3rds of the sample size of 1800. Interim review was conducted by a 3-member DSMB in January of 2010 and their recommendations were implemented.

ELIGIBILITY:
Inclusion Criteria:

* > 24 weeks, viable pregnancy, singleton or twins

Exclusion Criteria:

* No consent
* Contraindication to oxytocin
* Antepartum fetal demise
* Intrapartum use of concentrated oxytocin
* Planned cesarean
* DIC or coagulopathy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1798 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan T Tita, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Tita AT, Szychowski JM, Rouse DJ, Bean CM, Chapman V, Nothern A, Figueroa D, Quinn R, Andrews WW, Hauth JC. Higher-dose oxytocin and hemorrhage after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2012 Feb;119(2 Pt 1):293-300. doi: 10.1097/AOG.0b013e318242da74. PMID 22227638
- See also: PUBMED Abstract of Results — http://www.ncbi.nlm.nih.gov/pubmed/22227638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 1,798 women randomized.
Pre-assignment Details: At planned interim review (n=1,201), enrollment in the 40-unit group was stopped for futility and enrollment continued in the other groups.
Groups:
- Oxytocin 40 Units/500cc: Per DSMB recommendations, this intermediate arm was stopped Jan 2010.
Period: Overall Study
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Started | 659 | 481 | 658
Completed | 659 | 481 | 658
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc | Total
Number analyzed (Participants) | 659 | 481 | 658 | 1798
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 23.9 (5.4) | 23.9 (5.1) | 24.4 (5.5) | 24.2 (5.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 659 | 481 | 658 | 1798
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 143 | 97 | 156 | 396
  African American | 404 | 278 | 379 | 1061
  Hispanic | 106 | 101 | 120 | 327
  Other (not specified) | 6 | 5 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 659 | 481 | 658 | 1798

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Uterine Atony or Postpartum Hemorrhage Requiring Medical (Medication or Blood Transfusion), Surgical or Other Interventional Treatment
Description: the number of subjects with any treatment of uterineatony or hemorrhage.
Time Frame: baseline to discharge (2 - 3 days)
Measure: Number; unit: Participants
Groups:
- Oxytocin 10 Units/500cc; Oxytocin 80U/500cc: 1 dose only for prophylaxsis given over 1 hour
- Oxytocin 40 Units/500cc: Per DSMB recommendations, this intermediate arm was stopped Jan 2010.
  1 dose only for prophylaxsis given over 1 hour
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 659 | 481 | 658
Participants | 45 | 31 | 42

2. Primary Outcome: Women in Each Group With Risk Factors for Atony or Postpartum Hemorrhage
Description: In a secondary data analysis, a parsimonious set of independent risk factors for atony or postpartum hemorrhage was established: White, Hispanic, or Other (non-Black of African American) race/ethnicity, preeclampsia, or chorioamnionitus.
Time Frame: Initial hospital discharge (2-3 days)
Measure: Number; unit: participants
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 659 | 481 | 658
participants | 351 | 255 | 333

3. Secondary Outcome: Change in Pre- to Post-delivery Hematocrit (%)
Description: change in hematocrit from admission for delivery (baseline) to post-delivery (4 hours-1day postpartum depending on time of delivery)
Time Frame: During delivery hospitalization: Admission hematocrit - post-delivery hematocrit
Measure: Median (Inter-Quartile Range); unit: hematocrit difference (%)
Groups:
- Oxytocin 40 Units/500cc Over 1 Hour: Per DSMB recommendations, this intermediate arm was stopped Jan 2010.
Arm/Group | Oxytocin 10 Units/500cc Over 1 Hour | Oxytocin 40 Units/500cc Over 1 Hour | Oxytocin 80U/500cc Over 1 Hour
Number analyzed (Participants) | 659 | 481 | 658
hematocrit difference (%) | 4 [1 to 8] | 4 [1 to 8] | 4 [1 to 7]

4. Secondary Outcome: Number of Participants Experiencing Individual Treatment or Intervention in the Primary Outcome
Description: the number of individuals with each of the component treatments or individual outcomes in the primary composite.
Time Frame: prior to discharge
Measure: Number; unit: Participants
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 659 | 481 | 658
Participants
  Any Uterotonic | 45 | 30 | 40
  Blood Transfusion | 7 | 4 | 5
  Surgical | 0 | 0 | 1
  Other-Tamponade | 0 | 1 | 0
  Other-Arterial embolization | 1 | 0 | 1

5. Secondary Outcome: Number of Participants Experiencing Postpartum Hemorrhage (Clinical Estimate Greater Than 500cc)
Description: the number of individuals with a clinically estimated postpartum blood loss of 500cc or more
Time Frame: Initial hospital discharge (2-3 days)
Measure: Number; unit: Participants
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 659 | 481 | 658
Participants | 38 | 24 | 24

6. Secondary Outcome: Number of Subjects With Hospital Stays Greater Than 4 Days
Description: Number of individuals with prolonged hospitalization defined as 4 days or more prior to initial hospital discharge
Time Frame: Initial hospital discharge (2 days or more)
Measure: Number; unit: Participants
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 659 | 481 | 658
Participants | 116 | 95 | 109

7. Secondary Outcome: Number of Subjects Requiring Hypotension Warranting Pressor Agent or Fluid Bolus
Description: number of individuals with hypotension leading to administration of a fluid bolus or vasopressor agent (medication given to raise the blood pressure)
Time Frame: Initial hospital discharge (2-3 days or more)
Measure: Number; unit: Participants
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 659 | 481 | 658
Participants
  Pressor agent (medication given to increase BP) | 85 | 56 | 95
  Fluid bolus | 82 | 51 | 87

8. Primary Outcome: Risk to Using Increasing Doses of Oxytocin Based on Pre-specified Risk Factors
Description: The frequency of the primary study outcome is examined in a subgroup of 939 women with risk factors for atony or postpartum hemorrhage. These risk factors are identified as White, Hispanic, or Other (non-Black or African American) race/ethnicity, chorioamnionitis, and preeclampsia.
Time Frame: baseline to discharge (2-3 days)
Measure: Number; unit: participants
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Number analyzed (Participants) | 351 | 225 | 333
participants | 37 | 22 | 28
Statistical Analysis 1: Comparison: Oxytocin 10 Units/500cc vs Oxytocin 40 Units/500cc vs Oxytocin 80U/500cc; Test type: Superiority or Other; p = 0.670, ANCOVA; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.63 to 1.59]

ADVERSE EVENTS:
Arm/Group | Oxytocin 10 Units/500cc | Oxytocin 40 Units/500cc | Oxytocin 80U/500cc
Serious Adverse Events (participants affected / at risk) | 0/659 | 0/481 | 0/658
Other Adverse Events (participants affected / at risk) | 0/659 | 0/481 | 0/658

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of more than 60 days